CLINICAL TRIAL: NCT05224037
Title: Comparative Efficacy of Liver Fibrosis and Steatosis Assessment With Fibroscan and iLivTouch in Patients With Chronic Liver Diseases
Brief Title: Comparative Efficacy of Liver Fibrosis and Steatosis Assessment With Fibroscan and iLivTouch
Acronym: OGIG-01-22-LF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal State Budgetary Scientific Institution "Federal Research Centre of Nutrition, Biotechnology (Other)
Responsible Party: Principal Investigator, Sergey Morozov, Leading researcher, Federal State Budgetary Scientific Institution "Federal Research Centre of Nutrition, Biotechnology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FGMF-2022-0005
Record Dates: First submitted 2022-01-25; First posted 2022-02-04 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Chronic Liver Disease; Liver Fibrosis; Liver Steatoses
Keywords: ilivtouch; fibroscan; liver stiffness measurement; controlled attenuation parameter; non-alcoholic fatty liver disease; liver steatosis
MeSH Terms: conditions — Liver Cirrhosis; Fatty Liver; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): This is a single-arm study. All the participants will undergo examinations with 2 devices
  Interventions: Diagnostic Test: iLivTouch

INTERVENTIONS:
Diagnostic Test: iLivTouch — Eligible subjects will undergo liver stiffness and controlled attenuation parameters examination with two devices on the same day
  Other Names: FibroScan

SUMMARY:
This study is aimed to compare the results and operating characteristics of liver stiffness measurement with the use of Fibroscan (EchoSens, France) and iLivTouch (Wuxi Hisky Medical Technologies Co., China) in patients with chronic liver diseases.

DETAILED DESCRIPTION:
This is prospective comparative trial to assess diagnostic characteristics of non-invasive methods of liver fibrosis and steatosis assessment based on the measurement of liver stiffness. The null hypothesis is that novel device, iLivTouch FT100/FT200 and standard probe allows to obtain similar results of liver stiffness and controlled attenuation parameter compared to FibroScan 530 and probes M+ and XL+ in patients with chronic liver diseases. According to the study protocol, standard examination will be performed to eligible subjects on the same day with the use of both devices. At least 10 measurements will be performed with the use of each device to each subject after overnight fasting. The medians of liver stiffness and controlled attenuation parameter measurements, their interquartile range, success rate of measurements and related interpretations of the results (grades of liver fibrosis and steatosis) will be compared. To assess the variability of the results, demographic data (age, biological sex, ethnicity) will be collected; weight and height of the subjects will be measured on the day of examination. Medical history of the subjects will be examined to extract data, confirming the presence of chronic liver diseases and ensure eligibility.

ELIGIBILITY:
Inclusion Criteria:

* willingness to participate on the basis of the signed informed consent form;
* availability of the medical records

Exclusion Criteria:

* pregnancy and breastfeeding;
* narrow intercostal spaces making standard examination of the liver stiffness possible;
* extreme obesity, in cases when amount of the fat tissue in right lower part of chest makes impossible to perform measurements;
* ascites;
* focal lesions of the liver (including, but not limited to liver cancer or metastases of cancer regardless of their origin, parasitic invasions, cysts) in projection of the measurements;
* impossibility to perform evaluation with both devices due to any reasons;
* any health-related conditions of a subject that put him/her at risk in case the procedures required per study protocol are performed or making him/her ineligible on the discretion of the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Liver stiffness | Study day 1
  Single assessment (Median by at least 10 measurements) of the liver stiffness in kilo pascals will be performed during examination of the subject
Controlled attenuation parameter | Study day 1
  Single assessment (Median by at least 10 measurements) of the controlled attenuation parameter in kilo pascals will be performed during examination of the subject

SECONDARY OUTCOMES:
Interquartile range of liver stiffness | Study day 1
  Single assessment (interquartile range by at least 10 measurements) of the liver stiffness in kilo pascals will be performed during examination of the subject
Interquartile range of the controlled attenuation parameter | Study day 1
  Single assessment of interquartile range of the controlled attenuation parameter (by at least 10 measurements) in kilo pascals will be performed during examination of the subject
Success rate | Study day 1
  Success rate (a quotient of division of number of successful measurement on the total of number of measurements performed during examination of a subject) with iLivTouch and Fibroscan
Stage of liver fibrosis | Study day 1
  stage of liver fibrosis according to the liver stiffness and manufacturers instruction on the interpretation of the results of iLivTouch and FibroScan
Stage of steatosis of the liver | Study day 1
  stage of liver fibrosis according to the measurement of the controlled attenuation parameter obtained during examination of a subject and manufacturers instruction on the interpretation of the results of iLivTouch and FibroScan

CONTACTS AND LOCATIONS:
Overall Officials: Vasily Isakov, Professor, Study Chair — Federal State Budgetary Scientific Institution "Federal Research Centre of Nutrition, Biotechnology
Locations (1):
- Federal State Budgetary Scientific Institution "Federal Research Centre of Nutrition, Biotechnology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
depersonalised individual participants data may be shared upon reasonable request to the principal investigator after study completion
Supporting Information: Study Protocol, ICF, CSR
Time Frame: after study completion
Access Criteria: request to the investigator
URL: https://ion.ru